CLINICAL TRIAL: NCT00372905
Title: A Phase I/II Trial of Combined Weekly Bortezomib (VELCADE®) and Y-90-Ibritumomab Tiuxetan (Zevalin) in Patients With Relapsed or Refractory Follicular Lymphoma and Transformed Non-Hodgkin's Lymphoma
Brief Title: Phase I/II Trial of VELCADE Plus Zevalin in Patients With Relapsed or Refractory Follicular Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was closed permanently before the accrual goal was met due to slow accrual
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05H9; STU00004871 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma
Keywords: follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Bortezomib; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib, Ibritumomab tiuxetan, rituximab (Experimental): Induction therapy will last 28 days. Bortezomib will be given on days 1, 8, 15, and 22. Rituximab will be given on days 8 and 15 along with 111-indium-ibritumomab tiuxetan. During consolidation therapy, Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle for a maximum of 3 cycles. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
  Interventions: Drug: rituximab; Drug: bortezomib; Drug: Ibritumomab tiuxetan

INTERVENTIONS:
Drug: rituximab — Induction therapy will last 28 days. Bortezomib will be given on days 1, 8, 15, and 22. Rituximab will be given on days 8 and 15 along with 111-indium-ibritumomab tiuxetan. During consolidation therapy, Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle for a maximum of 3 cycles. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
  Other Names: Rituxan, IDEC-C2B8
Drug: bortezomib — Induction therapy will last 28 days. Bortezomib will be given on days 1, 8, 15, and 22. Rituximab will be given on days 8 and 15 along with 111-indium-ibritumomab tiuxetan. During consolidation therapy, Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle for a maximum of 3 cycles. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
  Other Names: Velcade
Drug: Ibritumomab tiuxetan — Induction therapy will last 28 days. Bortezomib will be given on days 1, 8, 15, and 22. Rituximab will be given on days 8 and 15 along with 111-indium-ibritumomab tiuxetan. During consolidation therapy, Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle for a maximum of 3 cycles. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
  Other Names: 111-indium-ibritumomab tiuxetan, Y-90-ibritumomab tiuxetan

SUMMARY:
Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Giving bortezomib together with rituximab and yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

This phase I/II trial is studying the side effects and best dose of bortezomib when given together with rituximab and yttrium Y 90 ibritumomab tiuxetan and to see how well they work in treating patients with relapsed or refractory follicular non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a phase I, dose-escalation study of bortezomib followed by a phase II study.

Phase I:

- Induction therapy: Patients receive bortezomib IV over 3-5 seconds on days 1, 8, 15, and 22, rituximab IV on days 8 and 15, and yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 15.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

- Consolidation therapy: Beginning 6-7 weeks after completing induction therapy, patients receive bortezomib IV over 3-5 seconds on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Phase II: Patients receive induction therapy and consolidation therapy as in phase I, with bortezomib administered at the MTD determined in phase I.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

A total of 24 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma
* CD20+ at time of diagnosis or subsequently
* More than 4 weeks since prior rituximab
* More than 3 weeks since prior anticancer therapy (6 weeks for nitrosourea or mitomycin C)
* More than 4 weeks since prior major surgery
* More than 2 weeks since prior investigational drugs

Exclusion Criteria:

* AIDS-related lymphoma
* History or evidence of CNS involvement
* Pregnant or nursing
* known HIV positivity
* serious medical or psychiatric illness that would preclude study participation
* myocardial infarction within the past 6 months
* congestive heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or ECG evidence of acute ischemia or active conduction system abnormalities
* known hypersensitivity to rituximab, bortezomib, boron, or mannitol
* prior autologous or allogeneic stem cell transplantation
* prior radioimmunoconjugate therapy or prior exposure to murine antibodies
* prior external-beam irradiation to > 25% of active bone marrow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-07-24 (Actual); Primary Completion 2010-06-22 (Actual); Study Completion 2013-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Winter, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on August 11, 2006 with an accrual goal of up to 24 patients. Accrual was suspended on September 9 2009 and reopened on November 30, 2009. The study was closed permanently on August 15, 2013 due to slow accrual with 18 patients enrolled and 17 patients treated on study.
Groups:
- Cohort 1: 1.0mg/m2 Bortezomib; Cohort 2: 1.3mg/m2 Bortezomib; Cohort 3: 1.6mg/m2 Bortezomib: Induction therapy will last one cycle of 28 days. Bortezomib will be given on days 1, 8, 15, and 22. 250mg/m2 of Rituximab will be given on days 8 and 15. 0.4mCi/kg of y-90-ibritumomab tiuxetan will be given on day 15.
  During induction therapy patients will receive either 1.0mg/m2, 1.3mg/m2, or 1.6mg/m2 of bortezomib as the study is designed as a 3+3 dose escalation of bortezomib to find the maximum tolerated dose.
  Consolidation therapy will last a maximum of 3 cycles and will start on day 71 (1 cycle = 28 days) During consolidation therapy, 1.6mg/m2 of Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
- Expansion Phase: 1.3mg/m2 Bortezomib: Induction therapy will last one cycle of 28 days. Bortezomib will be given on days 1, 8, 15, and 22. 250mg/m2 of Rituximab will be given on days 8 and 15. 0.4mCi/kg of y-90-ibritumomab tiuxetan will be given on day 15.
  During induction therapy patients will receive either 1.0mg/m2, 1.3mg/m2, or 1.6mg/m2 of bortezomib as the study is designed as a 3+3 dose escalation of bortezomib to find the maximum tolerated dose (MTD), or as the determined MTD in the expansion phase.
  Consolidation therapy will last a maximum of 3 cycles and will start on day 71 (1 cycle = 28 days) During consolidation therapy, 1.6mg/m2 of Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
Period: Cohort 1: Dose Level 1.0mg/m2
Arm/Group | Cohort 1: 1.0mg/m2 Bortezomib | Cohort 2: 1.3mg/m2 Bortezomib | Cohort 3: 1.6mg/m2 Bortezomib | Expansion Phase: 1.3mg/m2 Bortezomib
Started | 3 | 0 | 0 | 0
Registered to Study | 3 | 0 | 0 | 0
Treated 1 Cycle of Induction Therapy | 3 | 0 | 0 | 0
Completed 3 Cycles of Consolidation | 1 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 0 | 0 | 0
Period: Cohort 2: Dose Level 1.3mg/m2
Arm/Group | Cohort 1: 1.0mg/m2 Bortezomib | Cohort 2: 1.3mg/m2 Bortezomib | Cohort 3: 1.6mg/m2 Bortezomib | Expansion Phase: 1.3mg/m2 Bortezomib
Started | 0 | 3 | 0 | 0
Registered to Study | 0 | 3 | 0 | 0
Treated 1 Cycle of Induction Therapy | 0 | 3 | 0 | 0
Completed 3 Cycles of Consolidation | 0 | 3 | 0 | 0
Completed | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 3: Dose Level 1.6mg/m2
Arm/Group | Cohort 1: 1.0mg/m2 Bortezomib | Cohort 2: 1.3mg/m2 Bortezomib | Cohort 3: 1.6mg/m2 Bortezomib | Expansion Phase: 1.3mg/m2 Bortezomib
Started | 0 | 0 | 4 | 0
Registered | 0 | 0 | 4 | 0
Treated 1 Cycle of Induction Therapy | 0 | 0 | 3 | 0
Completed 3 Cycles of Consolidation | 0 | 0 | 1 | 0
Completed | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Expansion Phase at Dose 1.3mg/m2
Arm/Group | Cohort 1: 1.0mg/m2 Bortezomib | Cohort 2: 1.3mg/m2 Bortezomib | Cohort 3: 1.6mg/m2 Bortezomib | Expansion Phase: 1.3mg/m2 Bortezomib
Started | 0 | 0 | 0 | 8
Registration | 0 | 0 | 0 | 8
Treated 1 Cycle Induction Therapy | 0 | 0 | 0 | 8
Completed 3 Cycles of Consolidation | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2
Period: Follow up Until Relapse or Progression
Arm/Group | Cohort 1: 1.0mg/m2 Bortezomib | Cohort 2: 1.3mg/m2 Bortezomib | Cohort 3: 1.6mg/m2 Bortezomib | Expansion Phase: 1.3mg/m2 Bortezomib
Started | 3 (All patients that are treated on study move into the follow up phase at the completion of therapy.) | 3 | 3 | 8
Completed | 3 | 2 | 3 | 5
Not Completed | 0 | 1 | 0 | 3
Not completed — Study closed | 0 | 0 | 0 | 3
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bortezomib, Ibritumomab Tiuxetan, Rituximab: Induction therapy will last one cycle of 28 days. Bortezomib will be given on days 1, 8, 15, and 22. 250mg/m2 of Rituximab will be given on days 8 and 15. 0.4mCi/kg of y-90-ibritumomab tiuxetan will be given on day 15.
  During induction therapy patients will receive either 1.0mg/m2, 1.3mg/m2, or 1.6mg/m2 of bortezomib as the study is designed as a 3+3 dose escalation of bortezomib to find the maximum tolerated dose.
  Consolidation therapy will last a maximum of 3 cycles and will start on day 71 (1 cycle = 28 days) During consolidation therapy, 1.6mg/m2 of Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
Arm/Group | Bortezomib, Ibritumomab Tiuxetan, Rituximab
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Tolerability of Bortezomib Combined With Y-90-Ibritumomab Tiuxetan Determined by Number of Dose Limiting Toxicities in a Cohort.
Description: To determine the MTD using a 3+3 dose escalating design. There will be 3 dose cohorts:1.0mg/m2,1.3mg/m2 and1.6 mg/m2. 3 patients will be enrolled at dose of 1.0mg/m2 bortezomib. If no dose limiting toxicities (DLTs) are seen in the first 3 patients then dose will be escalated to next level and 3 patients will be treated at that dose level. If a DLT is seen at any dose, then 3 more patients will be enrolled at that dose level. If 1 patient out of 6, experience a DLT then MTD will be determined to be at this dose level. If 2 or more DLTs are seen in first 3 patients at that dose, then MTD will be one dose lower to the level where the DLTs were experienced.
  DLTs were defined using the National Cancer Institute Common Toxicity Criteria Version 3.0.
  DLTs=grade 3 nausea, vomiting, diarrhea or ileus more than 96h; grade 4 nausea, vomiting, diarrhea or ileus,neuropathic pain, peripheral sensory neuropathy, neutropenia, thrombocytopenia.
Time Frame: During induction therapy, the first 28 days of treatment.
Population: Patients enrolled in dose escalation cohorts 1, 2 and 3 analyzed for this outcome measure.
Measure: Number; unit: DLT
Arm/Group | Cohort 1: 1.0mg/m2 Bortezomib | Cohort 2: 1.3mg/m2 Bortezomib | Cohort 3: 1.6mg/m2 Bortezomib
Number analyzed (Participants) | 3 | 3 | 3
DLT | 0 | 0 | 2

2. Secondary Outcome: Number of Patients With Adverse Events Related to Treatment of Bortezomib Combined With Y-90-ibritumomab Tiuxetan
Description: To further explore the toxicity bortezomib combined with Y-90-ibritumomab tiuxetan by collecting data on adverse events (AE) reported by patient or collected lab results that are grade 3 or grade 4 that were determined to be at least possible related to any of the studies drugs.
  Toxicity will be collected on treatment days according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: At start of treatment on days 1, 8, 15, 22 of induction, days 36 and 50 of recovery, days 1, 8, 15 of consolidation cycles for up to 3 cycles and 4 weeks after the completion of treatment.
Population: Toxicity data for 9 patients enrolled in the dose escalating cohorts 1, 2 and 3 was collected and analyzed only. Data for the 3 cohorts are presented combined as the objective is to report grade 3 and 4 toxicities with this combination of drugs (dose of bortezomib is irrelevant)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1+ Cohort 2+ Cohort 3: Induction therapy will last one cycle of 28 days. Bortezomib will be given on days 1, 8, 15, and 22. 250mg/m2 of Rituximab will be given on days 8 and 15. 0.4mCi/kg of y-90-ibritumomab tiuxetan will be given on day 15.
  During induction therapy patients will receive either 1.0mg/m2, 1.3mg/m2, or 1.6mg/m2 of bortezomib as the study is designed as a 3+3 dose escalation of bortezomib to find the maximum tolerated dose.
  Consolidation therapy will last a maximum of 3 cycles and will start on day 71 (1 cycle = 28 days) During consolidation therapy, 1.6mg/m2 of Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
Arm/Group | Cohort 1+ Cohort 2+ Cohort 3
Number analyzed (Participants) | 9
Participants
  Leukopenia | 3
  Lymphopenia | 3
  Neutropenia | 5
  Thrombocytopenia | 4
  Cardiac | 1

3. Post Hoc Outcome: Overall Response Rate
Description: The overall response rate at the completion of treatment was defined as complete response plus partial response.
  Complete response (CR)=A post-treatment residual mass of any size is permitted as long as it is PET-negative and normalization of those biochemical abnormalities.
  Partial response (PR)=50% decrease in SPD of the six largest dominant nodes or nodal masses, no increase in the size of the other nodes, liver or spleen, and no new sites of disease.
  Stable disease=Failing to attain the criteria for PR or CR, but not fulfilling those for progressive disease.
  Progressive disease(PD)=At least a 50% increase from nadir in the SPD of any previously involved nodes or extranodal masses, or in a single involved node or extranodal mass, or the size of other lesions. Appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size.
Time Frame: At baseline, after induction cycle (1 cycle =28 days) and consolidation therapy of a maximum of 3 cycles (1cycle =28 days), up to approximately 6 months
Population: Data for first 9 patients enrolled in phase I dose escalation portion of the study were collected, analyzed and reported on. Cohort results for this outcome measure are combined as the objective was to determine the ORR of patients with this drug combination (dose was irrelevant)
Measure: Number; unit: percentage of patients
Arm/Group | Cohort 1+ Cohort 2+ Cohort 3
Number analyzed (Participants) | 9
percentage of patients | 89

4. Post Hoc Outcome: Median Progression Free Survival
Description: Median progression free survival (PFS) will be assessed by CT scans after induction therapy, consolidation therapy, every 3 months for the first year following treatment and every 6 months for the second year.
  Progressive disease is defined as the appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size or at least a 50% increase in the longest diameter of any single previously identified node or extranodal mass more than 1 cm in its short axis.
Time Frame: At start of treatment, at completion of induction therapy, at completion of consolidation therapy, every 3 months for 1 year, and every 6 months for 1 year
Population: The first 9 patients data that were enrolled in the phase I dose escalation portion were collected, analyzed and reported on. Cohort results for this outcome measure are combined as the objective was to determine the PFS of patients with this drug combination (dose was irrelevant)
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1+ Cohort 2+ Cohort 3
Number analyzed (Participants) | 9
Months | 6.5 [3 to 22.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) for the study were collected over a 5 year period. AEs for each patient were collected during treatment through 30 days post last treatment. Treatment consisted of one 28 day induction cycle followed by 71 day recovery period and then a maximum of 3 consolidation cycles each of 28 days.
Groups:
- Expansion Phase: 1.3mg/m2 Bortezomib: Induction therapy will last one cycle of 28 days. Bortezomib will be given on days 1, 8, 15, and 22. 250mg/m2 of Rituximab will be given on days 8 and 15. 0.4mCi/kg of y-90-ibritumomab tiuxetan will be given on day 15.
  During induction therapy patients will receive either 1.0mg/m2, 1.3mg/m2, or 1.6mg/m2 of bortezomib as the study is designed as a 3+3 dose escalation of bortezomib to find the maximum tolerated dose (MTD) or at the determined MTD in the expansion phase.
  Consolidation therapy will last a maximum of 3 cycles and will start on day 71 (1 cycle = 28 days) During consolidation therapy, 1.6mg/m2 of Bortezomib will be given intravenously on days 1, 8, and 15 of each cycle. Rituximab or Y-90-ibritumomab tiuxetan will not be given during consolidation therapy.
Arm/Group | Cohort 1: 1.0mg/m2 Bortezomib | Cohort 2: 1.3mg/m2 Bortezomib | Cohort 3: 1.6mg/m2 Bortezomib | Expansion Phase: 1.3mg/m2 Bortezomib
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 1.0mg/m2 Bortezomib (N=3) | Cohort 2: 1.3mg/m2 Bortezomib (N=3) | Cohort 3: 1.6mg/m2 Bortezomib (N=3) | Expansion Phase: 1.3mg/m2 Bortezomib (N=8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 1.0mg/m2 Bortezomib (N=3) | Cohort 2: 1.3mg/m2 Bortezomib (N=3) | Cohort 3: 1.6mg/m2 Bortezomib (N=3) | Expansion Phase: 1.3mg/m2 Bortezomib (N=8)
Otitis (non infectious) (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 1 | 2 | 3 | 4
Neutrophils (neutropenia) (Blood and lymphatic system disorders) | 3 | 2 | 2 | 2
Leukocytes (total white blood cells) (Blood and lymphatic system disorders) | 3 | 3 | 3 | 2
Lymphopenia (Blood and lymphatic system disorders) | 3 | 3 | 3 | 2
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 2 | 3 | 3 | 6
Hypertension (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac NOS (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 3 | 5
Fever (General disorders) | 0 | 0 | 0 | 1
Insomnia (General disorders) | 0 | 0 | 0 | 2
Sweating (General disorders) | 1 | 0 | 0 | 0
Weight loss (General disorders) | 0 | 0 | 0 | 1
Brusing (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritis/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Shingles (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hot flashes/flushes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Cavity - Root canal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 2 | 5
Distension/bloating abdominal (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Mucositis/stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Stomach upset (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hematoma (General disorders) | 0 | 1 | 0 | 0
Nose bleed (General disorders) | 0 | 1 | 0 | 0
Infection NOS (Infections and infestations) | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchus infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinus infection (Infections and infestations) | 1 | 0 | 0 | 3
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (skin rash) (Infections and infestations) | 1 | 0 | 1 | 0
Edema in limb(s) (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Edema of trunk/gential (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Edema of head/neck (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Alkaline phosphatase increase (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Transaminase (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
ALT increase (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Bilirubin increase (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Creatinine increase (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Calcium, serum high (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Calcium, serum low (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Glucose, serum high (Metabolism and nutrition disorders) | 2 | 3 | 1 | 2
Glucose, serum low (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Lactic acid dehydrogenase increase (LDH) (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Potassium, serum high (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Potassium, serum low (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Sodium, serum high (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Uric acid, serum high (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Neuropathy - motor (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy - sensory (Nervous system disorders) | 1 | 1 | 2 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1
Anxiety (Mood alteration) (Nervous system disorders) | 0 | 0 | 1 | 1
Agitation (Mood alteration) (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Fainting episode) (Nervous system disorders) | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Flank pain (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Mid thoracic pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 3
Pain in groin (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Shortness of breath (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study closed permanently due to slow accrual with only 17 patients treated on study. This was before the expected accrual goal of 24 patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes